CLINICAL TRIAL: NCT06361459
Title: Evaluation of the Influence of Stop Smoking to the Clinical and Radiological Outcome of Instrumented Neck and Back Surgery
Brief Title: Stop Smoking in Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Haga Hospital (Other); Alrijne Hospital (Other); Spaarne Gasthuis (Other)
Responsible Party: Principal Investigator, C.L.A.Vleggeert-Lankamp, MD MSc PhD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83858.058.12
Record Dates: First submitted 2024-01-04; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation
Keywords: smoking cessation, instrumented surgery, spondylodesis
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: three study groups: group that does not smoke, group that smokes and stops, group that smokes and does not stop
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stop smoking (Experimental): patients are stimulated to stop smoking, using the Sine Fuma program. after 4 weeks nicotine in urine will be tested. if stopped: planned for surgery. 4 weeks after surgery nicotine in urine is checked again. will be planned for surgery and evaluated
  Interventions: Behavioral: Stop smoking
- Continues smoking (Active Comparator): will be planned for surgery and evaluated
  Interventions: Behavioral: Stop smoking
- Does not smoke (No Intervention): will be planned for surgery and evaluated

INTERVENTIONS:
Behavioral: Stop smoking — Sine fuma program is offered. nicotine is checked in urine
  Arms: Continues smoking; Stop smoking

SUMMARY:
Patients that are subjected to a medium complex surgical intervention in neck (posterior) or lumbar spine (posterior) with instrumentation are motivated to stop smoking. The outcome data of patients that stop and that continue smoking will be compared. A group of non smokers is evaluated as a control group. Particularly clinical outcome is evaluated, as well as radiological outcome.

DETAILED DESCRIPTION:
Rationale: Optimizing outcomes of instrumented neck and back surgery Objective: To demonstrate that smoking cessation in the postoperative period has a positive impact on the clinical and radiological outcomes of instrumented spine surgery Study design: This is a multicenter observational cohort study with three groups of patients indicated to undergo moderately complex instrumented spinal surgery: a group of patients who continue to smoke is compared with a group who stop smoking in the peri-operative period of time. In addition, the results of a group of patients who do not smoke are recorded. Follow-up moments are baseline, 2, 6 and 12 months after surgery.

Study population: Patients between 18 and 75 years of age, who are candidates for moderately complex instrumented surgery of the neck or low back. Patients undergoing surgery for malignancy or trauma are excluded.

Intervention: If patients indicate that they are open to quitting smoking, they will be offered the SineFuma program. After 4 weeks, testing of nicotine in the urine will check whether smoking has actually stopped.

Study parameters: Primary outcome measure is the Oswestry Disability Index (low back) or the Neck Disability Index (neck). Furthermore, the VAS leg pain (or arm pain) and VAS back pain (or neck pain), the Hospital Anxiety and Depression Scale, the EuroQol and the patient's perceived recovery will be evaluated. The bony fusion will be assessed radiologically by CT at 6 and 12 months.

This is a multicenter observational cohort study adjusted for age and ASA score.

Evaluation moments: Patients will be asked to complete questionnaires at baseline and 2, 6 and 12 months after surgery. Patients who indicate that they have stopped smoking will be asked to submit a urine sample. For smokers who have to quit first, there is a second baseline measurement at the time they are scheduled for surgery. Data will be collected per center and brought together in the Data Coordination Center in Leiden (LUMC).

ELIGIBILITY:
Inclusion Criteria:

* candidates for moderately complex instrumented surgery of the neck or low back.

Exclusion Criteria:

* Patients undergoing surgery for malignancy or trauma are excluded.
* non Dutch speaking patients
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ODI or NDI | baseline, 2, 6 and 12 months post surgery
  Oswestry Disability Index (lumbar spine) or Neck Disability Index (neck surgery), ranging from 0 (best) to 100 (worst)

SECONDARY OUTCOMES:
VAS leg or arm pain | baseline, 2, 6 and 12 months post surgery
  VAS leg (lumbar spine) or VAS arm pain (neck surgery),ranging from 0 mm (best) to 100 mm (worst)
HADS | baseline, 2, 6 and 12 months post surgery
  Hospital Anxiety and Depression Scale, 2 scales ranging from 0 (best) to 18 (worst)
EuroQol | baseline, 2, 6 and 12 months post surgery
  quality of life, ranging from 0 (worst) to 1,0 (best)
perceived recovery | 2, 6 and 12 months post surgery
  perceived recovery in 7 grades ranging from 'completely recovered (= 1)' to 'much worse than I was before intervention (=7)'
radiological evaluation for fusion | 6 and 12 months after surgery
  CT scan to evaluate speed of fusion

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No